CLINICAL TRIAL: NCT04187469
Title: A Prospective, Randomized Controlled Study for the Efficacy and Safety of the Substitution of Pyrazinamide and Ethambutol With Moxifloxacin During the Intensive Phase of Treatment of Pulmonary Tuberculosis
Brief Title: Efficacy and Safety of Isoniazid, Rifampicin and Moxifloxacin for the Intensive Phase of Initial Therapy of PTB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Li Ding, Associate chief physician of infectious diseases, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.GRK.004
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Pulmonary Tuberculosis
Keywords: Pulmonary Tuberculosis; Anti-tuberculosis therapy; Intensive phase; Moxifloxacin; initial regimen
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Moxifloxacin; Isoniazid; Rifampin; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regimen 1: 2HRM/4HR (Experimental): Two month of chemotherapy with Moxifloxacin, Isoniazid and Rifampicin, followed by four month of Isoniazid and Rifampicin only.
  Interventions: Drug: Moxifloxacin, Isoniazid, Rifampicin
- Regimen 2: 2HRZE/4HR (control regimen) (Active Comparator): Two month of chemotherapy with Isoniazid, Rifampicin, Pyrazinamide and Ethambutol, followed by four month of Isoniazid and Rifampicin only.
  Interventions: Drug: Rifampicin,Isoniazid,Pyrazinamide,Ethambutol

INTERVENTIONS:
Drug: Moxifloxacin, Isoniazid, Rifampicin — Moxifloxacin 400 mg/day, Rifampicin ≤50 kg 450 mg/day > 50 kg 600 mg/day, Isoniazid 300 mg/day.
  All treatment is taken daily, for a duration of up to 6 months depending on treatment arm.
  Other Names: Avelox, Myambutol, Nydrazid, Rifampin, Rifadin
  Arms: Regimen 1: 2HRM/4HR
Drug: Rifampicin,Isoniazid,Pyrazinamide,Ethambutol — Rifampicin ≤50 kg 450 mg/day, >50 kg 600 mg/day, Isoniazid 300 mg/day, Pyrazinamide 1500mg/day, Ethambutol ≤50 kg or the elderly 750mg/day, >50 kg 1000mg/day.
  All treatment is taken daily, for a duration of up to 26 weeks depending on treatment arm.
  Other Names: Myambutol,Nydrazid,Rifampin,Rifadin
  Arms: Regimen 2: 2HRZE/4HR (control regimen)

SUMMARY:
This study aims to find an optimized initial regimen for pulmonary tuberculosis(PTB), evaluating the efficacy, safety and acceptability of isoniazid, rifampicin and moxifloxacin(HRM) for the intensive phase of initial therapy of PTB, compared with the standard initial regimen.

DETAILED DESCRIPTION:
The standard initial regimen for PTB consists of an initial 2-month intensive phase followed by a 4-month continuation phase. In the initial 2-month intensive phase, patients have to take four drugs-isoniazid, rifampin, pyrazinamide and ethambutol (HRZE) which might cause many adverse reactions. During the intensive phase, patients are prone to poor compliance due to adverse reactions, resulting in poor outcomes and drug-resistance. Therefore, it is necessary to optimize the regimen of intensive phase to improve patients' medication compliance, so as to avoid patients' treatment failure or drug resistance.

Moxifloxacin(M) has high antibacterial activity against both intracellular and extracellular Mycobacterium tuberculosis (Mtb) with few adverse reactions and is the most promising alternative to first-line anti-TB drugs. Isoniazid and rifampin have a strong bactericidal effect on both intracellular and extracellular Mtb. In the initial regimen for PTB, isoniazid and rifampin should be used throughout the whole process. They are the key drugs to ensure the curative effect and prevent recurrence, can not be easily replaced. But pyrazinamide and ethambutol just be used in the intensive phase. Pyrazinamide has the strongest killing effect on the intracellular Mtb and mainly exerts its antibacterial effect in the first two months of treatment. Ethambutol is a bacteriostatic drug, mainly effective for rapidly growing Mtb outside cells. They can lead to severe gastrointestinal reactions, liver damage, papilledema and other adverse reactions. So moxifloxacin might be an optional substitute for pyrazinamide and ethambutol.

This study will involve comparisons that are designed to assess the short-term efficacy, safety, relapse rate one year after drug withdrawal and patients' compliance when substituting moxifloxacin for pyrazinamide and ethambutol in the existing standard regimen. Patients selected for the study will be allocated to the trial group or the control group randomly. The control group will be given six months of a standard regimen(2HRZE/4HR). The trial group will be given a total of six months of treatment, with Substitution of pyrazinamide and ethambutol with moxifloxacin during the intensive phase(2HRM/4HR).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over, and an individual who completely bear the ability of civil actions.
* New cases of pulmonary tuberculosis. No previous anti-tuberculosis therapy or cumulatively taking anti-tuberculosis drugs for less than 1 month.
* Pulmonary tuberculosis patients with bacteriological diagnosis.

Exclusion Criteria:

* Suffering from tuberculous pleurisy.
* Patients with extrapulmonary tuberculosis.
* Renal insufficiency patients with creatinine clearance rate <30 ml/min.
* Abnormal liver function (ALT and/or AST and/or TBIL greater than 2 times the upper limit of normal) or decompensated cirrhosis.
* HIV-Ab positive.
* Psychiatric patients, or have a previous history of mental illness, or recently have obvious anxiety or depression and other mental abnormalities.
* Patients receiving immunosuppressive therapy.
* Pregnant or breast feeding.
* Diabetes.
* X-pert MTB/RIF test of sputum or alveolar lavage fluid showed that Mycobacterium tuberculosis was rifampin resistant.
* Moxifloxacin was used within 14 days before entering the group.
* Anti-tuberculosis treatment has been started and drugs are being taken before entering the group.
* QT interval extension > 480 ms.
* Combined with serious cardiovascular, liver, kidney, nervous system, blood system and other diseases or tumor diseases.
* Pulmonary lesions are widespread with respiratory insufficiency.
* Any other circumstances in which the anti-tuberculosis scheme of the experimental group or the control group cannot be selected for treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
The rate of adverse outcomes | 18 months (within one year of completion of therapy）
  Adverse outcomes: A sum of treatment failure and relapse.
  Treatment failure: A patient whose sputum smear or culture is positive at 5 months or later during treatment.
  Relapse: patients with successful treatment show one of the following conditions at any time point during the observation period of drug withdrawal: 1) Sputum or Bronchoalveolar lavage fluid(BALF)culture positive, 2) Sputum or BALF acid fast stain and/or Xpert positive with active PTB evidence in CT scan.

SECONDARY OUTCOMES:
The rate of Treatment success | the 2nd, 3rd, 5th and 6th months
  Treatment success: A sum of cured and completed treatment.
  Cure: A patient whose sputum smear or culture was positive at the beginning of the treatment but who was smear- or culture-negative in the last month of treatment and on at least one previous occasion.
  Treatment completed: A patient who completed treatment but who does not have a negative sputum smear or culture result in the last month of treatment and on at least one previous occasion.
The rate of sputum Mtb negative conversion | the 2nd, 3rd, 5th and 6th months
  Sputum Mtb negative conversion: two negative-culture results at different visits without an intervening positive result, or no sputum could be tested after once negative-culture.
The time of sputum Mtb negative conversion | the 2nd, 3rd, 5th and 6th months
  The first time of sputum Mtb negative conversion
Number of Patients With Adverse Events | 18 months (within one year of completion of therapy)
  The number of participants includes all patients who had adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Li Ding, M.D, Study Director — The Fifth Affiliated Hospital, Sun Yat-sen University; Yuanli Chen, M.Med, Principal Investigator — The Fifth Affiliated Hospital, Sun Yat-sen University; Xi Liu, M.D, Principal Investigator — The Fifth Affiliated Hospital, Sun Yat-sen University; JinYu Xia, M.Med, Principal Investigator — The Fifth Affiliated Hospital, Sun Yat-sen University; Zhongsi Hong, M.Med, Principal Investigator — The Fifth Affiliated Hospital, Sun Yat-sen University; Jian Liu, M.D, Principal Investigator — The Fifth Affiliated Hospital, Sun Yat-sen University; Minyi Lin, M.Med, Principal Investigator — The Fifth Affiliated Hospital, Sun Yat-sen University; Lisi Deng, M.Med, Principal Investigator — The Fifth Affiliated Hospital, Sun Yat-sen University; Lei Luo, Principal Investigator — The Fifth Affiliated Hospital, Sun Yat-sen University; Yayi Huang, Principal Investigator — The Fifth Affiliated Hospital, Sun Yat-sen University; Xiaoqing Luo, Principal Investigator — The Fifth Affiliated Hospital, Sun Yat-sen University; Yin Li, Principal Investigator — The Fifth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Fifth Affiliated Hospital Sun Yat-Sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tiberi S, du Plessis N, Walzl G, Vjecha MJ, Rao M, Ntoumi F, Mfinanga S, Kapata N, Mwaba P, McHugh TD, Ippolito G, Migliori GB, Maeurer MJ, Zumla A. Tuberculosis: progress and advances in development of new drugs, treatment regimens, and host-directed therapies. Lancet Infect Dis. 2018 Jul;18(7):e183-e198. doi: 10.1016/S1473-3099(18)30110-5. Epub 2018 Mar 23. PMID 29580819
- [Background] Lange C, Chesov D, Heyckendorf J, Leung CC, Udwadia Z, Dheda K. Drug-resistant tuberculosis: An update on disease burden, diagnosis and treatment. Respirology. 2018 Jul;23(7):656-673. doi: 10.1111/resp.13304. Epub 2018 Apr 11. PMID 29641838
- [Background] Pasipanodya JG, Gumbo T. A meta-analysis of self-administered vs directly observed therapy effect on microbiologic failure, relapse, and acquired drug resistance in tuberculosis patients. Clin Infect Dis. 2013 Jul;57(1):21-31. doi: 10.1093/cid/cit167. Epub 2013 Mar 13. PMID 23487389
- [Background] Egelund EF, Alsultan A, Peloquin CA. Optimizing the clinical pharmacology of tuberculosis medications. Clin Pharmacol Ther. 2015 Oct;98(4):387-93. doi: 10.1002/cpt.180. Epub 2015 Jul 22. PMID 26138226
- [Background] Pienaar E, Sarathy J, Prideaux B, Dietzold J, Dartois V, Kirschner DE, Linderman JJ. Comparing efficacies of moxifloxacin, levofloxacin and gatifloxacin in tuberculosis granulomas using a multi-scale systems pharmacology approach. PLoS Comput Biol. 2017 Aug 17;13(8):e1005650. doi: 10.1371/journal.pcbi.1005650. eCollection 2017 Aug. PMID 28817561
- [Background] Xu P, Chen H, Xu J, Wu M, Zhu X, Wang F, Chen S, Xu J. Moxifloxacin is an effective and safe candidate agent for tuberculosis treatment: a meta-analysis. Int J Infect Dis. 2017 Jul;60:35-41. doi: 10.1016/j.ijid.2017.05.003. Epub 2017 May 8. PMID 28495364
- [Background] Gillespie SH, Crook AM, McHugh TD, Mendel CM, Meredith SK, Murray SR, Pappas F, Phillips PP, Nunn AJ; REMoxTB Consortium. Four-month moxifloxacin-based regimens for drug-sensitive tuberculosis. N Engl J Med. 2014 Oct 23;371(17):1577-87. doi: 10.1056/NEJMoa1407426. Epub 2014 Sep 7. PMID 25196020
- [Background] Chakraborty S, Rhee KY. Tuberculosis Drug Development: History and Evolution of the Mechanism-Based Paradigm. Cold Spring Harb Perspect Med. 2015 Apr 15;5(8):a021147. doi: 10.1101/cshperspect.a021147. PMID 25877396
- See also: Definitions and reporting framework for tuberculosis — https://www.sogou.com/link?url=DSOYnZeCC_qzXHSs6m3Dx_BlXFNN_t5ZfNVVH3IkPP0cxjo-tKfxrn_Q9ViQ3mq_xcLO2TQn7Ac.